CLINICAL TRIAL: NCT03754816
Title: The Combination of PECS II Block and Parasternal Block Provide Useful Analgesia After Radical Mastectomy With Axillary Dissection and Implant Breast Reconstruction
Brief Title: The Combination of PECS II Block and Parasternal Block for Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Principal Investigator, San Salvatore Hospital of L'Aquila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0180910/16
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: PECS II block, parasternal block, analgesia
MeSH Terms: conditions — Breast Neoplasms; Agnosia | interventions — Levobupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The combination of PECS II and parasternal block performed by injecting Levobupivacaine 0.375% 40 ml, injected between minor and major pectoralis muscles, between minor and serratus muscles and between major and intercostal muscles
  Interventions: Procedure: PECS II and parasternal block; Drug: Levobupivacaine

INTERVENTIONS:
Procedure: PECS II and parasternal block — 10 ml of Levobupivacaine 0.375% injected between minor and major pectoralis muscles. 20 ml of Levobupivacaine 0.375% injected between minor and serratus muscles. 10 ml of Levobupivacaine 0.375% injected between major and intercostal muscles at II and IV intercostal space.
  Other Names: Pectoral nerve block II type and parasternal block
Drug: Levobupivacaine — Levobupivacaine
  Other Names: Locali anesthetic

SUMMARY:
The combination of PECS II and parasternal Block provides analgesia after radical mastectomy

DETAILED DESCRIPTION:
The cambionation of PECS II block and parasternal block

ELIGIBILITY:
Inclusion Criteria:

* ASA status patients:1,2 and 3
* patients undergoing to radical mastectomy with axillary dissection and breast-implant reconstruction

Exclusion Criteria:

* patients with allergy to local anesthetics
* ASA status patients: 4
* breast anatomy abnormalities
* neurological diseases
* septic conditions
* coagulopathies
* drug abuse history

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain: Numeric Rate Scale | 24 hours after surgery
  Postoperative pain evaluated with Numeric Rate Scale, from 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Intraoperative opiates | From start to the end of surgery
  Number of patients needing of equianalgesic mg of intraoperative morphine
Postoperative opiates | 24 hours after surgery
  Number of patients needing of equianalgesic mg of postoperative morphine
Side effects | 24 hours after surgery
  Number of patients with postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Petrucci, Principal Investigator — San Salvatore Academic Hospital of L'Aquila
Locations (1):
- San Salvatore Academic Hospital, Coppito, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No